CLINICAL TRIAL: NCT03237442
Title: Placebo-Controlled,Randomized,Double-blind Trial of Umbilical Cord Mesenchymal Stem Cells Injection for Ocular Corneal Burn
Brief Title: Umbilical Cord Mesenchymal Stem Cells Injection for Ocular Corneal Burn
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Saliai Stem Cell Science and Technology Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSCST-MSC-OCB-01
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Ocular Corneal Burn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental)
  Interventions: Biological: human umbilical cord mesenchymal stem cells
- group 2 (Active Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — human UC-MSCs: 0.2ml(about 2*10^6 cells) subconjunctival injection
  Arms: group 1
Biological: placebo — Saline injection
  Arms: group 2

SUMMARY:
Ocular chemical burn is one of the causes of vision loss in China, and there are no satisfactory treatment. Human umbilical cord mesenchymal stem cells(UC-MSCs) have the biological characteristics of self-renewal, immune regulation, multidirectional differentiation and tissue repair. Our preliminary research showed that in corneal alkali injury rabbits, the UC-MSCs can accelerated the cornea repair, inhibited angiogenesis. The aim of this study is to access the efficacy and safety of UC-MSCs in the treatment of corneal burn in human.

ELIGIBILITY:
Inclusion Criteria:

* must be ocular burns including chemically burned or the thermally burned;
* the subjects are willing to accept this research, and promise to coordinate with the researchers during the follow up period;
* the subjects should abide by the laws and rules of the study.

Exclusion Criteria:

* the visual acuity is blind in any of the eye;
* have corneal perforation or have the corneal perforation tendency;
* have been accepted surgery on eyeball after trauma;
* IOP>=25 mmHg even after antiglaucoma;
* have the history of other corneal disease or surgery;
* have the history of radiotherapy or surgery in the eyeball;
* associated with corneal ulcer or endoophthalmitis;
* uncontrolled hypertension(>=150/95 mmHg);
* abnormal liver and renal function;
* the pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
the percent of cornea perforation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China